CLINICAL TRIAL: NCT03310840
Title: A Observational Study on Ventilator-associated Pneumonia as a Risk for Nosocomial Infection in Mechanically Ventilated Neonates In NICU of Assiut University Children Hospital PROTOCOL OF THESIS Descriptive Study
Brief Title: A Study on Ventilator-associated Pneumonia as a Risk for Nosocomial Infection in Mechanically Ventilated Neonates In NICU of Assiut University Children Hospital (Nicu Eta)
Acronym: nicu eta
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd Elrhman Fawzy, M.B.B.CH resident doctor. principal investigator, Assiut University
Other Study IDs: PROTOCOL OF THESIS
Record Dates: First submitted 2017-09-25; First posted 2017-10-16 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Neonatal SEPSIS; Nosocomially Acquired Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Bro protein, Drosophila

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: others — others

SUMMARY:
Abstract

Background: Neonatal ventilator associated pneumonia (VAP) is a major hospital-acquired infection in acute care settings, associated with high mortality and poor outcome. VAP is considered a preventable infection if the risk factors are managed effectively. The purpose of this study is to evaluate prevalence of ventilator associated pneumonia, its causative organisms, its risk factors and outcome at our NICU.

This study used CDC guidelines for infant's ≤1 year old to diagnose neonatal VAP, in period from April 2018 to March 2019.

DETAILED DESCRIPTION:
Background:

Neonatal deaths represent third of the global burden of child mortality [1]. In Egypt, Infections such as pneumonia, meningitis, sepsis/septicemia and other infections account for 28% of deaths during the neonatal period, Survival cannot be achieved without substantial reductions in infection-specific neonatal mortality [2]. Neonatal sepsis is usually classified as early or late onset sepsis. Early sepsis occurs within the first 72 hours of birth and late neonatal sepsis occurs after 72 hours of birth. Early neonatal sepsis is associated with acquisition of microorganism from mother Late neonatal sepsis usually occurs due to the lack of aseptic working conditions [3]. The occurrence of late sepsis is considered an important indicator of quality of care. Mechanical ventilation is an essential, life-saving therapy for patients with critical illness and respiratory failure. These patients are at high risk for complications and poor outcomes, including death, Ventilator-associated pneumonia (VAP), Sepsis, pulmonary embolism, barotrauma, and pulmonary edema. Such complications can lead to longer duration of mechanical ventilation, longer stays in the intensive care unit (ICU) and hospital, increased healthcare costs, and increased risk of disability and death [4, 5]. Ventilator associated pneumonia (VAP) is defined as a nosocomial lower airway infection, i.e. pneumonia, in intubated patients with onset after 48 h or more of invasive mechanical ventilation [6]. VAP is usually caused by airway colonization by potential pathogens; Sources of airway colonization can be the patient's own flora, i.e., bacterial overgrowth in oral secretions, reflux and aspiration of gastric fluid or the patient's environment with its caretakers and equipment [7, 8].

Mechanically ventilated babies face a particular risk because artificial airways bypass the body's defenses against inhaled pathogens and offer new routes for non-air borne pathogens. Intubation associated lesions of pharynx and trachea lead to bacterial colonization by the deterioration of the swallowing reflex and the ciliary functions [9].VAP is one of the most frequently diagnosed nosocomial infections [10] and, after suspected early onset sepsis, second most reason for antibiotic intervention in Neonatal Intensive Care Unit (NICU) [11, 12].VAP incidence can be reduced by infection control measures such as VAP-prevention-bundles [13]. Regarding diagnosis of VAP episode requires a combination of radiological, clinical, and laboratory criteria. However Center for Disease Control and Prevention/ National Nosocomial Infection Surveillance (CDC/NNIS) criteria refers to infants younger than 1 year and do not define specific criteria for the newborn period in term or preterm infants. In spite of this lack of specificity, most studies of VAP performed in NICUs are based on these criteria [14].

Keywords: Newborn, Mechanical ventilation, ventilator-associated pneumonia, risk factors, causative organisms.

'Method's: Design: A prospective, observational cohort surveillance, was carried out at our Neonatal Intensive Care Unit (NICU) was done during a period from April 2018 to March 2019 to neonates who needed mechanical ventilation, reviewing data of diagnosis of neonates with ventilation associated pneumonia used .

Setting: Our NICU is a level III, part of a university-teaching hospital, receives referrals from the whole Upper Egypt. It has approximately 1450 case per year, approximately ~ 5 patients per day. It has approximately 450 case needs MV per year.

Patients:

Inclusion criteria:

All inborn and outborn neonates who were admitted to the our NICU during the April 2018- March 2019 were screened for study enrollment and were considered eligible if ventilated for more than 48 hours.

Exclusion criteria:

Neonates ventilated with Evidence of neonatal sepsis before ventilated. Meconium aspiration syndromes were excluded. Death within 48 hours of NICU admission.

• Neonates In our study were classified into two groups; i. Group A: cases with suspected VAP. ii. Group B: cases without VAP. Because up to this point we don't know the lab result and microbiology. The diagnosis should be based on all of the three items of radiologic signs, clinical signs and Symptoms and microbiological findings Cernada M et al [15].

Intervention:

* Medical records comprising charts, daily flow sheets, laboratory and radiographic reports were collected prospectively by the investigators.
* Neonates with suspected VAP in NICU: were diagnosed as VAP according to:

(Modified CDC guidelines for infants≤1 year old)[5,6,13].

All patient will be subjected to:

1. Full history taking:

   Including: Patient data, Perinatal history, Present history, Family history.
2. Full clinical examination:

   i. General physical assessment.
   1. Gestational age.
   2. Growth measurements.
   3. Vital data.
   4. General appearance. ii. Systems assessment.

   <!-- -->

   1. Neurological Examination.
   2. Respiratory Examination.
   3. Cardio-vascular Examination.
   4. Abdominal Examination. Then Monitoring of the ventilator settings, and fraction of inspired oxygen (FIO2).

   The clinical criteria for diagnosis; Worsening gas exchange: desaturations pulse oximetry less than 94%, increase ventilation demand,

   And at least three of the following Temperature instability Leukopenia (≤4000 WBC/mm3) or leukocytosis (>15,000 WBC/mm3) and left shift Band forms (10%) New onset of purulent sputum or change in character of sputum, or increased respiratory secretions Apnea, tachypnea, nasal flaring with retraction of chest wall or nasal flaring with grunting Wheezing, rales, or rhonchi
3. Investigation:

   1. Imaging study chest x-ray on admission& follow up, ultrasound, CT scan when indicated.
   2. Complete blood count, capillary blood gases. C) Septic screening

      1. Initial evaluation inflammatory mediator (C-reactive protein)
      2. Blood culture.
      3. Culture of bronchoalveolar lavage: aspirate for culture non-quantitative cultures after the third day hen weekly until extubation. Antibiotic sensitivity test will be done to all culture.

         We tried to compare the results of BAL versus blood culture in the diagnosis of VAP according to Cantey JB et al[12] ,aimed to intensive role of BAL.

         Microorganisms isolated from blood were compared with that isolated from BAL. According to results:

      <!-- -->

      1. Full agreement: when the same strain of organism has been isolated from the blood and endotracheal tube aspirate cultures,
      2. Partial agreement: when the organisms in the blood were found as one of the multiple isolates from the endotracheal tube,
      3. No agreement: when the organism was found in the endotracheal tube aspirate and blood was not the same,
4. Lines of treatment:

   * Initial (empirical) therapy is most often begun before a definite causative agent is identified.
   * Continuing therapy is based on culture and sensitivity results, clinical course

Ethical considerations:

The aim of the study was explained to each parents of the child before the beginning of the process. A written consent was obtained from those who welcomed to participate in the study. Privacy and confidentiality of all data were assured.

Statistical analysis:

The data were tested for normality using the Kolmogorov-Smirnov test and for homogeneity variances prior to further statistical analysis. Categorical variables were described by number and percent (N, %), where continuous variables described by mean and standard deviation (Mean, SD). Chi-square test used to compare between categorical variables where compare between continuous variables by t-test (One Way ANOVA). A two-tailed p < 0.05 was considered statistically significant. All analyses were performed with the IBM SPSS 20.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Characteristics: all cases All neonate admitted NICU of assiut University Children Hospital , who required endotracheal intubation and mechanical ventilation, regardless neonatal age.
* Target population, in details : all cases which develop neonatal sepsis on mechanically ventilate neonate admitted in NICU.of assiut university children hospital during the period from January 2018 to December 2018.

Exclusion Criteria

* meconium aspirated pneumonia .
* Neonates ventilated for infectious

Ages: 3 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: porotocal of thesis ;
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
mechanical ventilation accused to be risk factor for nosocomial infection in neonate . | from april 2018 to march 2019
  to determine incidence and prevalence of neonatal sepsis on mechanically ventilated neonate

SECONDARY OUTCOMES:
value of Surveillance program | from april 2018 to march 2018
  serial endo tracheal aspirate ever three day to predict neonatal sepsis and type of organisms causing sepsis in ventilated neonate,antibiotic proper usage

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University NICU of Children Hospital, Asyut, Egypt